CLINICAL TRIAL: NCT03504254
Title: Plasticity of Chronically Compressive Spinal Cord After Surgical Decompression - A fMRI Study
Brief Title: A fMRI Study of Compressive Spinal Cord
Acronym: CSM Plasticity
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW12-468
Record Dates: First submitted 2017-12-05; First posted 2018-04-20 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2019-09

CONDITIONS: Orthopedic Disorder of Spine; Neurologic Disorder
Keywords: cervical spondylotic myelopathy; diffusion tensor imaging; functional magnetic resonance imaging
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CSM: A total of 50 CM patients requiring surgical decompression will be recruited. The inclusion criteria are a clinical diagnosis of CM including the signs of corticospinal lesions together with the appropriate radiographic findings. Patients with acute spinal cord injuries, prior spinal intervention or claustrophobia will be excluded.
  Interventions: Diagnostic Test: MRI examination

INTERVENTIONS:
Diagnostic Test: MRI examination — Three kinds of MRI techniques will be used in this study. These are (1) axial T1-weighted (T1WI) and T2-weighted imaging (T2WI), UTE MRI, (2) BOLD-based fMRI, and (3) diffusion tensor imaging (DTI).

SUMMARY:
Cervical myelopathy (CM), a chronically compressive spinal cord lesion, is the most common cause of non-traumatic paraparesis/quadriparesis among the elderly. Hong Kong is facing a heavy social economic burden from CM with the rapidly aging population. Surgical decompression is considered as the mainstay of the treatment for CM patients to relieve their symptoms and signs. Yet the surgical outcome is not always satisfactory. There is a pressing need for understanding the exact mechanism of surgical decompression on the recovery of myelopathic cord in order to improve the prognosis of CM patients in near future.This project will evaluate neuronal activities and axon regeneration by longitudinally monitoring at time zero, 3 and 6 month after the surgery in CM patients using UTE, BOLD-fMRI and DTI, and to investigate the relationship of preoperative neuronal activities of myelopathic cord with axon regeneration.

DETAILED DESCRIPTION:
This study aims to monitor the structural and functional changes of chronically compressed spinal cords longitudinally after surgical decompression in vivo. Three kinds of MRI techniques will be used in this study. These are (1) axial T1-weighted (T1WI) and T2-weighted imaging (T2WI), UTE MRI, (2) BOLD-based fMRI, and (3) diffusion tensor imaging (DTI). To quantitatively investigate the structural deficits, T1/T2 MRIs will delineate the gross morphology of the spinal cord, CSF, and surrounding anatomical structures, while DTI will quantify the fiber orientation and integrity within the spinal cord. BOLD-based functional MRIs will assess the local hemodynamic changes and neuron activities in response to the motor or sensory stimulation along the C3 to C8 spinal nerve levels. The MRI evaluations will be applied to the same cervical myelopathy (CM) patient before surgery and 3 and 6 months post-surgery, when clinical recovery reaches a plateau9. Clinical examination will include neurological evaluation, Japanese Orthopaedic Association (JOA) scoring assessment, and clinical electrophysiological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are a clinical diagnosis of CM including the signs of corticospinal lesion/s together with the appropriate radiographic findings.

Exclusion Criteria:

* Patients with acute spinal cord injuries, prior spinal intervention or claustrophobia will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 CM patients requiring surgical decompression will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-01-11 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
DTI indics | Change between Enrollment and one year after surgery.
  The mean diffusivities and fractional anisotropy will be measured in the DTI

SECONDARY OUTCOMES:
fMRI connextivity | Change between Enrollment and one year after surgery.
  Functional connectivity will be examined by calculating the averaged correlation coefficient of all regions of interest (ROIs) in gray matters.

CONTACTS AND LOCATIONS:
Locations (1):
- The university of Hong Kong, Hong Kong, Hong Kong